CLINICAL TRIAL: NCT00424710
Title: Phase I Study of Ranibizumab Injection for Polypoidal Choroidal Vasculopathy (PEARL)
Brief Title: Ranibizumab for Polypoidal Choroidal Vasculopathy (PCV)
Acronym: PEARL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hawaii Pacific Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Gregg T. Kokame, MD, Medical Director, The Retina Center at Pali Momi, Hawaii Pacific Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF3934s
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: choroidal neovascularization
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy; Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm study (Other): Single arm study:
  Drug: ranibizumab intravitreal injection liquid, 0.5 mg ranibizumab intravitreally, once a month for 1 year
  Interventions: Drug: ranibizumab intravitreal injection

INTERVENTIONS:
Drug: ranibizumab intravitreal injection — liquid, 0.5 mg ranibizumab intravitreally, once a month for 1 year

SUMMARY:
This is a 12 month study of monthly injections of ranibizumab in subjects with polypoidal choroidal vasculopathy as diagnosed by fluoresceins/indocyanine green (FA/ICG) angiography.

DETAILED DESCRIPTION:
Previous treatment in subjects is allowed as long as appropriate washout period has elapsed. Patients will be followed by 4M ETDRS vision testing as well as scheduled OCT, ICG, FA and Fundus Photography.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent and comply with study assessment for the duration of one year
* Age >= 25 years
* Polypoidal Choroidal Vasculopathy as noted on fluorescein and ICG angiography: active leakage, active bleeding or recent decrease in vision
* BCVA using ETDRS 20/32 to 20/400

Exclusion Criteria:

* Any history of previous vitrectomy
* Previous cataract or ocular surgery within 2 months of day 0
* Active intraocular inflammation in the study eye
* Active infections conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Participation with another investigational drug within the past 30 days
* Prior sodium pegaptanib, verteporfin photodynamic therapy, intravitreal steroids, or bevacizumab within 30 days of study entry
* Blood pressure >180/110 (use of antihypertensives is allowed as long as hypertension can be controlled and is stable)
* Pregnancy

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Efficacy Measured by the proportion of subjects who lose fewer than 15 letters in visual acuity at 6 and 12 month compared with baseline | 1 year
Safety and Tolerability as measured by the recording and observations of adverse effects of study treatment | 1 Year

SECONDARY OUTCOMES:
Efficacy as measured by the mean change from baseline in VA at 6 and 12 months | 1 Year
Efficacy as measured by the proportion of subjects who lose less than 5 letters of vision at month 6 and 12 | 1 Year
Efficacy as mean change from baseline at 6 to 12 months in decreasing subretinal hemorrhage or subretinal exudates via fundus photographs and fundus exams | 1 Year
Efficacy as proportion of subjects with a decrease in size of the polypoidal vessels from PCV at Mo 6 and 12 as assessed by FA and ICG Angiography | 1 Year
Efficacy as proportion of subjects with a decrease in macular edema as measured by OCT in central or paracentral fields from baseline month 6 and month 12. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Gregg T Kokame, MD, Principal Investigator — The Retina Center at Pali Momi
Locations (2):
- United States (2):
  - Retina Consultants of Hawaii, Honolulu, Hawaii
  - The Retina Center at Pali Momi, ‘Aiea, Hawaii

REFERENCES:
- [Result] Kokame GT, Yeung L, Lai JC. Continuous anti-VEGF treatment with ranibizumab for polypoidal choroidal vasculopathy: 6-month results. Br J Ophthalmol. 2010 Mar;94(3):297-301. doi: 10.1136/bjo.2008.150029. Epub 2009 Sep 1. PMID 19726427